CLINICAL TRIAL: NCT06064136
Title: Psoas Tenotomy Under Ultrasound
Acronym: TEPSe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-AOIP-07
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with ilio-psoas conflict and having a tenotomy indication (Experimental)
  Interventions: Procedure: Psoas tenotomy under ultrasound

INTERVENTIONS:
Procedure: Psoas tenotomy under ultrasound — Tenotomy of the ilio-psoas tendon under ultrasound is performed using an ultrasound machine, a 3 mm Acufex hook blade and a specific kit usually used for guided vertebroplasty and which allows the introduction of the Acufex hook blade atraumatically (foam end). The patient, under general anesthesia, is placed in supine position with the hip extending from 15 to 20°.

SUMMARY:
The ilio-psoas conflict is a commonly accepted complication after total hip replacement, often linked to a mispositioning of the acetabular prosthetic component that conflicts with the ilio-psoas tendon. To correct these pains, a psoas tenotomy can be proposed. The results proven by the literature are very satisfactory. Psoas tenotomy is performed endoscopically, arthroscopically, or more rarely open.

The contribution of echo surgery allows to limit the scar ransom but also to free itself from a complex infrastructure to the operating room including an arthroscopy column and an intraoperative fluoroscopy for a conventional tenotomy, This also saves procedural and installation time.

No studies to date have described ultrasound-assisted psoas tenotomy Yhe investigators conducted a cadaveric study of the feasibility of psoas tenotomy under ultrasound that confirms the feasibility of this technique and the safety of the gesture for the surrounding anatomical structures.

The objectives of this study are to assess the feasibility, pain and functional outcomes of ultrasound-assisted psoas tenotomy in patients with ilio-psoas conflict after total hip replacement.

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years of age or older
* Indication of psoas tenotomy for ilio-psoas conflict after total hip replacement
* Signature of the written informed consent form by the patient
* Affiliation to a French health insurance scheme or equivalent

Non Inclusion criteria:

* Vulnerable people: pregnant or breast-feeding women (patients will undergo a pregnancy test: urinary test), adult under guardianship or deprived of freedom.
* Allergies to local anesthetics
* Patient on anticoagulant or antiplatelet agents
* Contraindication to surgery
* Refusal of patient involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the success rate of this new ultrasound-guided ilio-psoas tendon tenotomy technique | 3 weeks post-operative
  The success of this new ultrasound-guided ilio-psoas tendon tenotomy technique will be assessed by the disappearance of the ilio-psoas conflict after surgery. This criterion will be measured at the first control consultation

SECONDARY OUTCOMES:
Evaluate the new ultrasound-guided ilio-psoas tendon tenotomy technique compared to standard practice on pain experienced by the patient | Pre-operative, 3 hours, 1 day, 3 weeks, 6 weeks, 3 and 6 months post-operative
  The pain felt by the patient will be collected using a numerical scale from 0 to 10 before surgery, 3 hours after surgery, the day after surgery, then 3 weeks, 6 weeks, 3 months and 6 months after surgery. Zero '0', means that the patient has no pain ; '10', means that the patient has extreme pain. The non-inferiority limit is set at 1.5 on the pain EVA scale
Evaluate the Oxford Hip Score | At baseline, 3 weeks, 6 weeks, 3 and 6 months post-operative
  The Oxford Hip Score is a questionnaire that assesses pain and hip function of patients who have undergone total hip replacement surgery. Patient should reflect on their pain and functional abilities on the previous 4 weeks. The questionnaire is divided into 2 domains (pain and function), each domain being composed of 6 questions. For each question, 5 answers are possible, each with a score of 0 to 4 (None = 4, Minimal = 3, Slight = 2, Moderate = 1, Severe = 0). The total score ranges from 0 (most severe symptoms) to 48 (no symptoms).
Evaluate the Harris Hip Score | At baseline, 3 weeks, 6 weeks, 3 and 6 months post-operative
  The Harris Hip Score assess the results of hip surgery. It is composed of 10 questions divided into 4 domains (pain, function without deformation and amplitude of movements). A score is assigned to each response. The total score varies from 0 to 100. The higher the score, the better the results and the less dysfunctional the patient
Evaluation the Postel and Merle Aubigne score | At baseline, 3 weeks, 6 weeks, 3 and 6 months post-operative
  the Postel and Merle Aubigne score measures pain, joint mobility and walking. For each question, 6 answers are possible, each one having a score of 0 to 6. The total score varies from 0 to 18, 18 indicating a perfect hip
Evaluate the technical difficulty of surgical procedure | the day after surgery
  The technical difficulty of surgical procedure will be assessed using a 4-point Likert scale: on the day of the operation, the surgeon will have to answer the question "What was the difficulty experienced by you in the operation?". He may answer by: Very difficult, difficult, moderately difficult or easy.
Evaluate the operative time | the day of surgery
  The operative time will be expressed in minutes between skin incision and skin closure
Evaluate the installation time | the day of surgery
  The installation time will be expressed in minutes between the end of intubation and the beginning of the brush
Evaluate the total blood loss | in the month before surgery and the day after surgery
  Total blood loss will be calculated according to the ostheo formula, including pre-operative (in the month preceding the surgery) and post-operative (the day after surgery) hematocrit values. This measure makes it possible to accurately assess the hidden blood losses related to the hematic extravasation
Evaluate the length of hospital stay | the day after surgery
  The length of hospital stay will be expressed in hours, between the entry and the discharge of the patient
Evaluate the scarring after surgery | 6 weeks post-operative
  The scarring after surgery will be evaluated at 6 weeks after surgery using a subjective scar satisfaction score (4-point Likert scale), transmitted by the patient himself. The patient will have to answer the question "Are you satisfied with your scar?". He can answer: Very satisfied, satisfied, dissatisfied or very dissatisfied.
Evaluate the impact of the patient's quality of life | At baseline, 6 weeks, 3 and 6 months post-operative
  Quality of life will be evaluated using the EuroQol five-dimension questionnaire (EQ-5D-5L), at inclusion, 6 weeks, 3 and 6 months after surgery.The EQ-5D-5L comprises a descriptive system and a visual analogue scale (VAS). The descriptive system is composed of five health dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) with 5 levels of health (no problems, slight problems, moderate problems, severe problems and extreme problems). For each of the 5 dimensions, the participant's answer is converted to a number between 1 and 5, expressing the health state reported. The responses are combined to produce a five-digit number describing the participant's health status which is converted to a utility value from the country specific value set. The French EQ-5D-5L value set has utility between -0.530 (health condition worse than death) and 1 (best possible health). The VAS records the self-rated health status on a graduated scale from 0 to 100.
Evaluate the patient satisfaction with the results of the operation | 3 weeks, 6 weeks, 3 and 6 months post-operative
  Patient satisfaction will be assessed at 3 weeks, 6 weeks, 3 months and 6 months post-surgery using a 4-point Likert scale. To do this, the patient will have to answer the question: "Are you satisfied with the results of your surgery?". They can answer with: very satisfied, satisfied, dissatisfied, or very dissatisfied.
Evaluate the subjective value of the hip | at baseline, 3 weeks, 6 weeks, 3 and 6 months post-operative
  The subjective value of the hip will be assessed at inclusion, 3 weeks, 6 weeks, 3 months and 6 months after surgery by the patient himself. By answering the question "What then is the overall percentage value of your hip if a completely normal hip equals 100%?" , the patient should assess his hip on a scale of 0 to 100, 100 corresponding to a perfect hip.
Evaluate the forgotten hip sensation | 3 weeks, 6 weeks, 3 and 6 months post-operative
  The forgotten hip sensation will be assessed by the patient himself at 3 weeks, 6 weeks, 3 months and 6 months after surgery by answering the question "Have you forgotten your hip?". The patient can answer yes or no.
Evaluate the Forgotten Hip score. | at baseline, 6 weeks, 3 and 6 months post-operative
  The forgotten hip score will be assessed at inclusion, 6 weeks, 3 and 6 months after surgery. The score is composed of 12 questions assessing the degree of forgetfulness. For each question, the patient may respond with never, almost never, rarely, sometimes, often.
Evaluate the early (< 90 days) and late (> 90 days) surgical complications related to surgery | During 6 months after surgery
  Early complications (< 90 days after surgery) and late complications (> 90 days after surgery) will be sought the day after surgery and throughout the follow-up period. They will be classified as major (infections at the surgical site or medical complications increasing the length of hospitalization) or minor according to the series of the literature
Evaluate the rate of patient requiring a stay in a rehabilitation center | During 6 months after surgery
  The number of patients requiring rehabilitation will be collected for the duration of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No